CLINICAL TRIAL: NCT02752438
Title: Rescue High Frequency Oscillatory Ventilation in Newborns Who Do Not Respond to Conventional Ventilation
Acronym: RescueHFO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Collaborators: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other); Etlik Zubeyde Hanim Womens (Unknown); Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other); Gazi University (Other); Istanbul Medeniyet University (Other); Dr. Behcet Uz Children's Hospital (Other); Celal Bayar University (Other); Special Metro Hospital (Other); Konya Meram State Hospital (Other); Inonu University (Other)
Responsible Party: Principal Investigator, Omer Erdeve, Prof. Dr. Omer Erdeve, Ankara University
Other Study IDs: RescueHFO
Record Dates: First submitted 2016-04-23; First posted 2016-04-27 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Acute Mechanical Ventilatory Failure
Keywords: high frequency oscillatory ventilation; rescue; newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Survived: Patients who are treated with HFOV at least for 4 h in case of unresponse to conventional ventilation and survived.
  Interventions: Device: HFOV
- Death: Patients who are treated with HFOV at least for 4 h in case of unresponse to conventional ventilation but died.
  Interventions: Device: HFOV

INTERVENTIONS:
Device: HFOV — HFOV is a kind of respiratory support with a rate higher than physiological but with lesser volume.

SUMMARY:
Although High Frequency Oscillatory Ventilation (HFOV) has been used in case of unresponsive to conventional mechanical ventilation both in children and newborns, there is no data on its success and the factors that affect its success in the literature.

DETAILED DESCRIPTION:
Although High Frequency Oscillatory Ventilation (HFOV) has been used in case of unresponsive to conventional mechanical ventilation both in children and newborns, there is no data on its success and the factors that affect its success in the literature.

The aim of the study is to define the factors that affect the success of HFOV in newborns who do not respond to conventional mechanical ventilation through an online registry among neonatal intensive care units in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* patients switched to HFOV in case of unresponse to conventional ventilation
* stay on HFOV for at least 4 h

Exclusion Criteria:

* any congenital anomaly
* HFOV duration less then 4 h

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns with respiratory insufficiency in spite of conventional mechanical ventilation are candidates for the study. When the patient is switched to HFOV for rescue respiratory support, he/she will be followed and registered to online registry system.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Survival | 3 months

SECONDARY OUTCOMES:
Cut-off gestational age for survival | 3 months
Cut-off birthweight for survival | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Omer Erdeve, Principal Investigator — Ankara University
Locations (1):
- Ankara University Children's Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared.